CLINICAL TRIAL: NCT01660828
Title: The Effect of Remote Ischemic Preconditioning on Plasma Troponin I Appearance After a Standardized Cycling Test in Healthy Volunteers
Brief Title: Exercise Test and Cardiac Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EXTROP2
Record Dates: First submitted 2012-07-23; First posted 2012-08-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Disease
Keywords: Exercise induced (high sensitive) troponin release; Ischemia reperfusion injury; Remote ischemic preconditioning
MeSH Terms: conditions — Cardiovascular Diseases; Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive cycling test preceded by RIPC (Active Comparator): Intensive cycling test preceded by a RIPC protocol.
  Interventions: Other: remote ischemic preconditioning (RIPC)
- No intervention/ RIPC (No Intervention): Intensive cycling test not preceded by a RIPC protocol.

INTERVENTIONS:
Other: remote ischemic preconditioning (RIPC) — RIPC protocol which consist of three 5-min cycles of bilateral forearm ischemia
  Arms: Intensive cycling test preceded by RIPC

SUMMARY:
Strenuous exercise in apparent healthy individuals increases plasma (high sensitive) troponin levels. The underlying mechanism is not yet elucidated, but could be explained by changes due to a mismatch in oxygen demand and supply that mimic those of ischemia and reperfusion injury. If the mechanism underlying the troponin release during exercise is similar to that of ischemia reperfusion injury (IRI), than it should be susceptible to remote ischemic preconditioning (RIPC) as RIPC is a well validated technique to reduce IRI. To test this hypothesis healthy volunteers underwent a strenuous exercise test with or without preceding RIPC.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-45 year
* willing to sign informed consent
* healthy

Exclusion Criteria:

* hypertension (systolic blood pressure >140 mmHg or diastolic blood pressure > 90 mmHg)
* any cardiovascular abnormality in past medical history, physical examination or ECG, including QTc interval
* drug abuse
* alcohol abuse (> 3 units/day)
* smoking during the last 2 years
* BMI >30 kg/m2
* inability to perform bicycle test
* the presence of an absolute or relative contra-indication for exercise (table 2 in protocol)
* the presence of diabetes (fasting glucose > 6.9 mmol/L, non-fasting glucose >11.0 mmol/L; if non-fasting glucose is > 6.9 mmol/L, blood glucose measurement will be repeated in fasting condition and should then not exceed 6.9 mmol/L)
* total cholesterol in blood 6.6 mmol/L or higher

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
serum level of high sensitive troponin at several timepoints | timepoints t= baseline, 0, 1, 2, 3,4 and 8 hours after finishing exercise
  serum level of high sensitive troponin in response to intensive exercise test with or without RIPC at several timepoints

CONTACTS AND LOCATIONS:
Overall Officials: G. Rongen, MD, PhD, Principal Investigator — Radboud University Nijmegen Medial Centre
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands